CLINICAL TRIAL: NCT01222507
Title: Processing Speed as an Objective Measure of Tinnitus
Acronym: BST
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Posit Science Corporation (Industry)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine, Washington University School of Medicine
Other Study IDs: 10-0829
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-09

CONDITIONS: Tinnitus
Keywords: tinnitus; cognition; brain processing speed; Brain Fitness Program; Posit Science
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Speed Test: 60 subjects who complete 60 Second Brain Game and Brain Speed Test

SUMMARY:
The overall purpose of this research is to assess whether both the "60 second Brain Game" and the "Brain Speed Test" computer-based programs can be used as assessment tools for objectively defining the severity of the functional impact of tinnitus.

DETAILED DESCRIPTION:
This cross-sectional study aims to assess for deficits in brain processing speed and attention (two cognitive domains whose deficits have been implicated in tinnitus) with the use of the "Brain Speed Test".

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18 and 80.
* Participants must have subjective, unilateral or bilateral, non-pulsatile tinnitus of 6-months duration or longer.
* Participants must be able to read, write and speak using the English language.
* Participants must be able to provide informed consent.

Exclusion Criteria:

* Participants with tinnitus related to Workman's Compensation Claim or other litigation-related situations.
* Participants with active diagnoses of any acute or chronic brain-related neurological conditions that alter normal brain anatomy or function including Parkinson's disease, Multiple Sclerosis, Alzheimer's Disease, cerebral infarcts, traumatic brain injury, history of brain tumor(s), epilepsy, or dementia.
* Participants with tinnitus related to retrocochlear lesions, cochlear implants, or other known anatomic/structural lesions of the brain, skull-base, temporal bone or ear.
* Participants unable to hear the highest volume of the computer-based objective assessments.
* Any medications that may affect or alter cognition including but not limited to sedatives, hypnotics, narcotics, or opiates.
* Any medical condition the PI determines would compromise the safety of the participant or complicate the interpretation of the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tinnitus subjects recruited from speciality clinic and community at large.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Piccirillo, MD, Principal Investigator — Washington Unieversity
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Washington University ENT and Audiology Clinics, as well as from Washington Univerity Volunteers for Health recruitment enhancement core.
Pre-assignment Details: 2 subjects failed to meet inclusion/exclusion criteria after signing consent form.
Groups:
- Brain Speed Test (BST): 60 subjects who complete 60 Second Brain Game and Brain Speed Test
Period: Overall Study
Arm/Group | Brain Speed Test (BST)
Started | 62
Completed | 60
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brain Speed Test
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Brain Speed Test
Description: This test involves the presentation of two consecutive high or low-frequency sound sweeps that requires the participant to correctly identify the order of presentation of the sound sweeps. Correct identification of the sound sweeps requires intact brain processing speed and attention. Scores are presented relative to age-matched controls used in validating the test. The normative data for the controls for this test will be provided by Posit Science® to the PI.
Time Frame: Initial study visit
Population: The number of subjects who completed the study according to protocol.
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- Brain Processing Speed: Brain Speed Test is measured through Brain Speed Test, and the results are transformed to z-scores based on normal population data.Z-score is calculated by subtracting the raw score (x) from the mean of the population (µ) which is then divided by the standard deviation of the population.
Arm/Group | Brain Processing Speed
Number analyzed (Participants) | 60
units on a scale | -0.28 [-0.58 to 0.10]

ADVERSE EVENTS:
Time Frame: One time assessment
Arm/Group | Brain Speed Test
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No